CLINICAL TRIAL: NCT06772064
Title: Efficacy of Rifaximin in Patients With Small Intestinal Bacterial Overgrowth Presenting With Abdominal Bloating: An Exploratory Study.
Brief Title: Efficacy of Rifaximin in Patients With Small Intestinal Bacterial Overgrowth Presenting With Abdominal Bloating.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiuli Zuo (Other)
Responsible Party: Sponsor-Investigator, Xiuli Zuo, Professor, Director of gastroenterology department of Qilu hospital., Shandong University
Organization: Shandong University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-202408-061-1
Record Dates: First submitted 2024-12-22; First posted 2025-01-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: SIBO
Keywords: SIBO; Abdominal bloating; Rifaximin
MeSH Terms: interventions — Rifaximin; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy group (No Intervention): The healthy group met the inclusion and exclusion criteria, and stool samples were retained for microflora analysis as control.
- Patient group (Experimental): Patients were required to collect stool samples and score a psychopsychological questionnaire. After enrollment, patients were given Rifaximin dry suspension 0.4g bid for 2 weeks. During the medication period, patients' drug consumption and adverse reactions were recorded through diary cards. After 2 weeks of medication, diary cards and outer packaging of drugs were collected, and case report forms were supplemented. Stool samples were collected again, anxiety and depression scale scores were performed, and clinical symptom changes were recorded. The breath test was reviewed 1 month after the end of the medication, and follow-up was conducted 3 months and 6 months after the end of the medication.
  Interventions: Drug: Rifaximin (drug)

INTERVENTIONS:
Drug: Rifaximin (drug) — Rifaximin 0.4g bid for 2 weeks
  Arms: Patient group

SUMMARY:
Abdominal bloating is a common clinical symptom in the digestive system, with obscure origins and complex mechanisms. Its etiology can be attributed to organic diseases and various Functional Gastrointestinal Disorders (FGIDs). In recent years, the roles of Small Intestinal Bacterial Overgrowth (SIBO), Oral-Cecal Transit Time (OCTT), and gut microbiota dysbiosis in Functional Abdominal Bloating/Distention (FAB/D) have garnered increasing attention. Currently, there is a lack of diagnostic tests and effective treatment measures for patients with bloating. The hydrogen/methane breath test is a safe, economical, and non-invasive examination recommended for diagnosing SIBO. Rifaximin, an antibiotic that acts exclusively in the intestines, has been widely validated for its efficacy in SIBO and in patients with SIBO co-occurring with Irritable Bowel Syndrome (IBS). However, research on the role of SIBO in the production of bloating symptoms and the extent to which rifaximin treatment of SIBO alleviates symptoms in clinical bloating patients is still lacking. This study aims to investigate the efficacy of rifaximin in patients with SIBO who primarily present with bloating. Exploring clinical treatment options for bloating provides a reference for its management. Furthermore, questionnaires on psychiatric symptoms and fecal microbiota analysis for patients with bloating-type SIBO can help clarify the etiology of bloating, offering a basis for the etiological treatment of bloating patients in the next steps.

DETAILED DESCRIPTION:
The study enrolled subjects who primarily complained of abdominal bloating, and underwent breath testing, along with healthy volunteers. Study participants were required to meet the inclusion criteria, not meet the exclusion criteria, and sign an informed consent form. After enrollment, they completed a case report form. Basic demographic information of the study participants, results of routine laboratory tests, clinical characteristics related to symptoms, results and values of breath test, and other data were recorded. Patients were required to provide stool samples and conduct psychiatric questionnaire scoring, and the healthy control group was also required to provide stool samples. After enrollment, patients took rifaximin dry suspension at a dosage of 0.4 g twice a day for two weeks, recording medication intake and adverse reactions through a diary card during the medication period. Two weeks after the end of the medication, the diary cards and medication packaging were collected, and the case report forms were supplemented. Stool samples were taken again, and anxiety and depression scale scores were recorded to document changes in clinical symptoms. One month after the end of the medication, patients were required to undergo a repeat breath test, and follow-ups for changes in abdominal bloating symptoms were conducted three and six months after the end of the medication .

ELIGIBILITY:
Healthy Group

Inclusion Criteria:

1. Age between 18 and 70 years, both genders included.
2. No special gastrointestinal discomfort such as bloating or abdominal pain, regular bowel movements, and normal stool characteristics.
3. Negative hydrogen/methane breath test.

Exclusion Criteria:

1. Pregnant or lactating women.
2. History of gastrointestinal malignancy or gastrointestinal surgery.
3. Past diagnosis or suspicion of lactose intolerance.
4. Confirmed extra-digestive system diseases such as urinary system (chronic kidney disease, etc.), immune system (scleroderma, etc.), nervous system (Parkinson's, etc.), endocrine system (diabetes, etc.).
5. Abnormalities in professional anxiety and depression symptom rating scales.
6. Use of antibiotics, probiotics within two weeks, endoscopic examination, or use of prokinetics, secretagogues, antifoaming agents, antispasmodics, opioids, antidepressants within one week.
7. Those who cannot or are unwilling to sign an informed consent form.

Patient Group:

Inclusion Criteria:

1. Age between 18 and 70 years, both genders included.
2. Chief complaints of abdominal bloating and/or distension; outpatients with abdominal bloating and/or distension more prominent than other symptoms.
3. Positive hydrogen/methane breath test.

Exclusion Criteria:

1. Pregnant or lactating women.
2. History of gastrointestinal malignancy or gastrointestinal surgery.
3. Past diagnosis or suspicion of lactose intolerance.
4. Confirmed extra-digestive system diseases such as urinary system (chronic kidney disease, etc.), immune system (scleroderma, etc.), nervous system (Parkinson's, etc.), endocrine system (diabetes, etc.).
5. Moderate to severe abnormalities in professional anxiety and depression symptom rating scales.
6. Use of antibiotics, probiotics within two weeks, endoscopic examination, or use of prokinetics, secretagogues, antifoaming agents, antispasmodics, opioids, antidepressants within one week.
7. Those who cannot or are unwilling to sign an informed consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Negative conversion rate of hydrogen and methane breath testing | Up to 1 week after hydrogen and methane breath testing
  Negative conversion rate of hydrogen and methane breath testing in patients treated with rifaximin.

SECONDARY OUTCOMES:
Symptom remission rate | During the administration period, 1 month after the end of the administration, 3 months and 6 months of follow-up
  Symptom remission rate in patients treated with rifaximin

OTHER OUTCOMES:
Changes of fecal flora (16 S Sequence Analysis). | Immediately collect fecal before and after taking rifaximin.
  Changes of fecal flora before and after rifaximin administration.
The difference of fecal flora between patients and normal population (16 S Sequence Analysis). | Test immediately after collection of stool sample.
Psychopsychological questionnaire score | Collect the questionnaire and rate it immediately.
  Self-rating depression scale (SDS): minimum value: 20; maximum value:100;The dividing line between normal and anxious patients is 50 points, with higher scores indicating more severe anxiety.
  Self-Rating Anxiety Scale (SAS): minimum value: 20; maximum value:100; In the Chinese population, the dividing line between normal and depressed people is 53 points, with higher scores indicating more severe depression.
  Hamilton Anxiety Scale (HAMA):minimum value: 0; maximum value:56; The dividing line between normal and anxious patients is 7 points, with higher scores indicating more severe anxiety.
  Hamilton Depression Scale (HAMD): minimum value: 0; maximum value: 96; the dividing line between normal and depressed people is 8 points, with higher scores indicating more severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No